CLINICAL TRIAL: NCT00337740
Title: Randomized Study Comparing Ligation With Propranolol for Primary Prophylaxis of Variceal Bleeding in Candidates for Liver Transplantation
Brief Title: Banding Versus Propranolol for Primary Prophylaxis of Variceal Bleeding
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: From the interim analysis resulted that more than 1000 patients were required to demonstrate a significant difference between the 2 treatments.
Sponsor: University of Padova (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TCPSVECE/9/01PD
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2012-04-23 (Estimated); Status verified 2006-09

CONDITIONS: Liver Cirrhosis; Esophageal Varices
MeSH Terms: conditions — Liver Cirrhosis; Esophageal and Gastric Varices | interventions — Propranolol

INTERVENTIONS:
Procedure: endoscopic variceal banding
Drug: propranolol

SUMMARY:
Whether beta-blockers or banding is the best therapy for primary prophylaxis of variceal bleeding is subject to debate. A randomized comparison between the two treatments was performed in candidates for liver transplantation. Patients with Child B and C cirrhosis with high risk varices and no previous variceal bleeding are randomized to propranolol or variceal bleeding. Primary end point is variceal bleeding

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis
* child pugh>=B7
* studied for transplantation
* age between 18 an 65 ys
* no previous bleeding from varices
* signed informed consent

Exclusion Criteria:

* esophageal varices less than F2 blue
* gastric varices
* previous variceal surgical or radiological or endoscopical treatment
* hepatocarcinoma
* portal vein thrombosis
* severe heart, respiratory or renal failure
* contraindications to betablockers
* treatment with nitrates, calcium antagonist or anti-arhythmic drugs that can not be suspended
* Pregnancy
* neoplasias
* non cooperation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)

PRIMARY OUTCOMES:
variceal bleeding

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Norberto, prof, M.D., Principal Investigator — University of Padova, Department of Surgical and Gastroenterological Sciences, 1st Surgical Clinic; Umberto Cillo, prof. M.D., Principal Investigator — University of Padova, Department of Surgical and Gastroenterological Sciences, 1st Surgical Clinic; Francesco Grigoletto, prof, M.D., Study Director — Biostatistic and Epidemiology Unit, Department of Enviromental Medicine and Public Health, University of Padova, Italy; Davide D'Amico, prof, MD, Study Chair — Padova University, Department of Surgical and Gastroenterological Sciences, 1st Surgical Clinic
Locations (1):
- Clinica Chirurgica 1^, Policlinico Universitario, Via Giustiniani 2, Padua, Italy